CLINICAL TRIAL: NCT01152372
Title: Experimental Medicine Study to Validate the Modified Glucose Disposal Test in Healthy Subjects and Subjects With Type 2 Diabetes
Brief Title: Experimental Study to Validate the Modified Glucose Disposal Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MB122-003
Record Dates: First submitted 2010-06-16; First posted 2010-06-29 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Other): Beta cell function by frequently sampled intravenous glucose tolerance test
  Interventions: Procedure: Insulin, glucose and staple isotopes
- Arm 2 (Other): Modified glucose disposal test assessment of insulin sensitivity, endogenous glucose production and insulin secretion
  Interventions: Procedure: Insulin, glucose and staple isotopes
- Arm 3 (Other): Endogenous glucose production and insulin sensitivity by isotope dilution and isoglycemic, heperinsulinemic clamp
  Interventions: Procedure: Insulin, glucose and staple isotopes

INTERVENTIONS:
Procedure: Insulin, glucose and staple isotopes

SUMMARY:
Evaluate the modified GDT as a measure of key metabolic characteristics in healthy subjects and those with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes
* Clinically healthy
* Drug naive or on a stable dose of metformin monotherapy and/or a secretagogue

Exclusion Criteria:

* Type 1 Diabetes
* History of significant heart disease.
* Bariatric surgery
* Exposure to fibrates, thiazolidinediones, insulin, exenatide, pramlintide or DPP-IV inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Glucose (labeled and unlabeled), insulin and c-peptide will be measured to calculate insulin sensitivity, endogenous glucose production and insulin secretion | within 24 hours

SECONDARY OUTCOMES:
Characterize the patterns of intermediate metabolites in healthy subjects and subjects with type 2 diabetes mellitus | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Profil Institute For Clinical Research, Inc. (Picr), Chula Vista, California, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx